CLINICAL TRIAL: NCT05885503
Title: A Phase III, Multicenter, Randomized, Double-blind, Active Controlled Trial of RC28-E Intravitreal Injection in Subjects With Diabetic Macular Edema
Brief Title: Efficacy and Safety of RC28-E Versus Aflibercept in Diabetic Macular Edema
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28C005
Record Dates: First submitted 2023-05-19; First posted 2023-06-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC-28E (Experimental): RC-28E 2.0 mg will be initially intravitreal injected (IVT) 5 times at 4 week intervals from week 0 to week 16, then every 8 weeks until week 48.
  Interventions: Biological: RC-28E
- Aflibercept (Active Comparator): Aflibercept 2.0mg will be received IVT once every 4 weeks for 5 consecutive times from week 0 to week 16, then once every 8 weeks till week 48.
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Biological: RC-28E — Ophthalmic solution for intravitreal injection administered as a 2.0mg/50 μL per dose.
  Arms: RC-28E
Biological: Aflibercept — Ophthalmic solution for intravitreal injection administered as a 2.0mg/50 μL per dose.
  Arms: Aflibercept

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of RC28-E compared with Aflibercept in subjects with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosed with type I or type II diabetes mellitus.
* Hemoglobin A1c (HBA1c) of less than or equal to (≤) 10% within 2 months prior to Day 1.
* Ability and willingness to undertake all scheduled visits and assessments.
* The study eye must meet the following requirements:

  * macular thickening secondary to diabetic macular edema (DME) involving the center of the fovea.
  * decreased visual acuity attributable primarily to DME, the best corrected visual acuity (BCVA) 19 or more letters, 78 letters or less.

Exclusion Criteria:

* The study eye with high risk of proliferative diabetic retinopathy.
* The macular edema of the study eye is mainly caused by other diseases or factors other than DME.
* Treatment with panretinal photocoagulation or macular laser within 3 months prior to Day 1 to the study eye.
* Administration of IVT any other anti-VEGF drugs in the study eye within 3 months and/or in the other eye within 7 days prior to Day 1.
* Any intraocular long-acting or sustained release corticosteroid treatment (e.g., dexamethasone intravitreal implant) in the study eye within 6 months prior to Day 1.
* Active intraocular or periocular infection or active intraocular inflammation in either eye.
* The study eye with poorly controlled glaucoma.
* A history of idiopathic or autoimmune related uveitis in either eye.
* History of stroke (cerebrovascular accident) or myocardial infarction within 6 months prior to Day 1.
* Uncontrolled blood pressure, defined as a systolic value greater than (>)180 millimeters of mercury (mmHg) and/or a diastolic value >100 mmHg while a patient is at rest.
* Currently pregnant or breastfeeding, or intend to become pregnant during the study.
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision in the study eye.
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than DME in the study eye.
* Other protocol-specified inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in BCVA at Week 52 | Baseline, week 52
  BCVA=best-corrected visual acuity; Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a starting distance of 4 meters

SECONDARY OUTCOMES:
Average change in BCVA from baseline over the period week 40 through week 52 | Baseline, weeks 40, 44, 48 and 52
  For each subject, this endpoint is defined as the average of the changes from baseline to weeks 40, 44, 48 and 52
Change from baseline in BCVA over time | Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  BCVA will be assessed at each visit
Proportion of patients gaining >15, >10, >5, or >0 letters in BCVA from baseline at Week 52 | Baseline, week 52
  Proportion of patients of gaining 4 types of letter counting in BCVA, respectively
Proportion of patients avoiding a loss of >15, >10, >5, or >0 letters in BCVA from baseline at Week 52 | Baseline, week 52
  Proportion of patients of reducing 4 types of letter counting in BCVA, respectively
Change from baseline in CST at Week 52 | Baseline, week 52
  CST=central subfield thickness
Mean change from baseline in CST over a period of week 40 through week 52 | Baseline, weeks 40, 44, 48 and 52.
  CST=central subfield thickness
Change from baseline in CST over time | Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
  The change of CST will be assessed from baseline to 52 weeks by every 4 week intervals
Proportion of patients with absence of intraretinal fluid at Week 52 | Baseline, week 52
  Proportion of patients whose intraretinal fluid are completely improved
Proportion of patients with absence of subretinal fluid at Week 52 | Baseline, week 52
  Proportion of patients whose subretinal fluid are completely improved
Proportion of patients with absence of intraretinal fluid and subretinal fluid at Week 52 | Baseline, week 52
  Proportion of patients whose intraretinal fluid and subretinal fluid are both completely improved
Proportion of patients with a >2-step or>3-step DRS worsening from baseline on ETDRS DRSS at Week 52 | Baseline, week 52
  DRSS=Diabetic Retinopathy Severity Scale
Proportion of patients who develop new PDR or high risk PDR at Week 52 | Baseline, week 52
  PDR=proliferative diabetic retinopathy
Incidence and severity of ocular adverse events and non-ocular adverse events | 0~52 weeks
  during the study
Plasma concentration of RC28-E over time | Baseline, weeks 16, 36 and 48
  during the study
Presence of ADAs during the study relative to the presence of ADAs at baseline | Baseline, weeks 12, 24, 36 and 52
  during the study

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided